CLINICAL TRIAL: NCT01958879
Title: Treatment of Temporomandibular Disorder
Brief Title: Efficacy of Arthrocentesis by Injection of Ringer With or Without Corticosteroid in Treatment of Internal Derangement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, OMFS, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2013-10-05; First posted 2013-10-09 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Temporomandibular Joint Dysfunction; Pain; Arthrocentesis
Keywords: internal derangement,arthrocentesis,corticosteroid
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ringer with corticosteroid (Experimental): Intra-articular irrigation was performed under local anesthesia with subcutaneous injection of 1%lidocaine solution (0.6 to 0.9 mL anaesthetic solution )was injected to block the auriculotemporal nerve. Then the skin on the TMJ was penetrated with a 21-gauge needle at the articular fossa followed by the injection of 3 mL Ringer solution to distend the joint space, pumping it in and out repeatedly. Another 21-gauge needle was inserted into the distended compartment in the area of the articular eminence, and the superior joint space was irrigated with 200 mL Ringer solution, allowing a free flow through the first needle in the both groups .In this group patients received 1mg dexamethasone after finishing the irrigation .
  Interventions: Drug: ringer with corticosteroid
- Ringer with out corticosteroid (Placebo Comparator): Intra-articular irrigation was performed under local anesthesia with subcutaneous injection of 1%lidocaine solution (0.6 to 0.9 mL anaesthetic solution )was injected to block the auriculotemporal nerve. Then the skin on the TMJ was penetrated with a 21-gauge needle at the articular fossa followed by the injection of 3 mL Ringer solution to distend the joint space, pumping it in and out repeatedly. Another 21-gauge needle was inserted into the distended compartment in the area of the articular eminence, and the superior joint space was irrigated with 200 mL Ringer solution, allowing a free flow through the first needle in the both groups
  Interventions: Drug: ringer without corticosteroid

INTERVENTIONS:
Drug: ringer with corticosteroid — 200 mL Ringer solution+1mg dexamethasone after finishing the irrigation
  Arms: ringer with corticosteroid
Drug: ringer without corticosteroid — 200 mL Ringer solution
  Arms: Ringer with out corticosteroid

SUMMARY:
The study aims to evaluate effectiveness of ringer injection with or without corticosteroid during arthrocentesis of the temporomandibular joint in the treatment of internal derangement of the temporomandibular joint (TMJ).

DETAILED DESCRIPTION:
This prospective clinical study was approved by Local ethical committee and written informed consent will be obtained before the trial starts. Criteria for selection of the patients was based on history and clinical findings characteristic of internal derangement. All these patients were initially treated with NSAIDS for 1 week and occlusal splints for 1 month had failed to respond to these conservative treatments. The patients with systemic problems which affect bone and joints,psychological problems ,history of maxillofacial fractures and orthognathic surgery were excluded from the study. A total of 60 patients with TMJ internal derangement with failed conservative management, were subjected to TMJ arthrocentesis. All arthrocentesis were performed by the same maxillofacial surgeon. Subjects were randomly allocated into two groups (30 cases in each group). Subjects in the group 1 received irrigation with Ringer solution and in the group 2 ,subjects underwent irrigation with Ringer solution with corticosteroid (Dexamethasone ) .Two examiners evaluated Temporomandibular disorder's signs ( mouth opening,click , crepitus and pain) before, one month and 6 months after arthrocentesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical findings characteristic of internal derangement(clicking and joint pain lasting for more than 6 months) unilaterally or bilaterally and history of previous conservative drug therapy (NSAIDs and Muscle relaxant ),splint therapy and physiotherapy without improvement.
* Patients of both sexes between 15 to 80 year's old
* Patients who are willing for evaluation in 1 and 6 months after arthrocentesis
* Patients who are provided written consent form

Exclusion Criteria:

* Patient had systemic problems which affect bone and joints disease
* Patient with psychological problems
* Patient with history of maxillofacial fractures and orthognathic
* Patients who can not continue the study for private or social reasons

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
pain | 6 months
  Pain will be assessed preoperatively and again at 1 and 6 months using a visual analogue scale

SECONDARY OUTCOMES:
function | 6 months
  Mouth opening was measured as the maximum interincisal distance in millimeters using a scale

CONTACTS AND LOCATIONS:
Overall Officials: Reza Tabrizi, DMD, Study Chair — SUMS; Reza Tabrizi, DMD, Study Director — SUMS; Touba Karagah, DMD, Principal Investigator — SUMS
Locations (1):
- Shiraz university of medical sciences, Shiraz, Iran